CLINICAL TRIAL: NCT05031741
Title: A Pilot Intervention to Reduce Adolescent Sexual and Mental Health Disparities by Increasing Access to Telemedicine and Mobile Care (AccessKCTeen)
Brief Title: Reducing Adolescent Sexual and Mental Health Disparities by Increasing Access to Telemedicine and Mobile Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Melissa Miller, Principal Investigator, Physician, Children's Mercy Hospital Kansas City
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00001900
Record Dates: First submitted 2021-08-20; First posted 2021-09-02 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Health Care Utilization
Keywords: teen program; sexual health; mental health; AccessKCTeen
MeSH Terms: conditions — Patient Acceptance of Health Care; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: We will assign participants a Telemedicine or In-person Mobile unit card as they enroll in the study at events. Teens with a telemedicine card will get education exposure to telemedicine with a video and an ipad that demonstrates a pretend telehealth visit. Teens with an In-person mobile unit card will have the opportunity to learn how a health visit can be done on the unit with a health care provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telemedicine (Experimental): Teens who are randomly assigned a telemedicine card will have exposure to a pretend telemedicine visit equipped with an iPad and telehealth provider on the other end. The study team will demonstrate how a teen can acquire sexual and reproductive health as well as mental health care through telemedicine from their own home or private space.
  Interventions: Other: Peer Leader Model
- In-person Mobile Unit (Experimental): Teens who are randomly assigned a in-person mobile unit card will have exposure to a pretend mobile unit visit equipped with a healthcare provider. The study team will demonstrate how a teen can acquire sexual and reproductive health as well as mental health care on the mobile unit.
  Interventions: Other: Peer Leader Model

INTERVENTIONS:
Other: Peer Leader Model — Teens will have an opportunity to interact with established peer leaders that are a part of the AccessKCTeen program. These leaders will receive a baseline training of their role, sexual and mental health. They will also receive health education and engage with a peer liason via text messages throughout the study.

SUMMARY:
Investigators will attend a series of community outreach events that provide/demonstrate telemedicine and the Children's Mercy Mobile Unit which is equipped to provide direct patient care. Investigators will engage up to 12 teen peer leaders to encourage healthcare-seeking behaviors and mobilize their social networks to attend outreach events. At all events, the mobile unit will be available for teens to (a) demonstrate the mobile unit and telehealth experience; (b) learn about Sexual and Reproductive Health/Mental Health (SRH/MH) and local care resources; (c) register for future telemedicine care; (d) acquire free over-the-counter emergency contraception, condoms, and pregnancy tests.

DETAILED DESCRIPTION:
AccessKCTeen is a pilot clinical outreach program that uses Children Mercy's Mobile Unit and Telemedicine to demonstrate and increase access to SRH and MH. AccessKCTeen intends to focus on these central activities:

1. Education based on a peer-leader model: In collaboration with community-based partners, investigators will identify and train approximately 12 peer leaders in disseminating information and resources for MH/SRH to their social networks. Peer leaders may disseminate information in the form of sharing curated online resources or mobilizing friends to attend live educational events. Peer leaders will also help connect their friends to resources by spreading information and encouraging friends to attend CM mobile unit demonstrations. Investigators will use text messaging to engage peers in these educational events and share general health resources.
2. Mobile Unit and Telemedicine Demonstration Events: The mobile unit will be present at community events to demonstrate how in-person care could work on the unit as well as how telemedicine works. Investigators will answer questions and help adolescents get registered for telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Telemedicine or In-person Mobile unit arms: Aged 14-18 years old and Attended a Mobile Unit Demonstration
* Peer leaders: At least 14 years old

Exclusion Criteria:

* Telemedicine or In-person Mobile unit arms: Younger than 14 years old, 19 years of age or older, did not attend a Mobile Unit Demonstration, does not speak/understand English
* Peer leaders: Younger than 14 years old

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Uptake of any Sexual and Reproductive/Mental Health Care in past 30 days | one month
  Look at the uptake frequency in Sexual and Mental health care among participants within 30 days of baseline and educational interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Miller, MD, Principal Investigator — Children's Mercy; Emily Hurley, PhD, Principal Investigator — Children's Mercy
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States